CLINICAL TRIAL: NCT07353554
Title: Application Study of 68Ga-NOTA-BCMA Nanoantibody Imaging in Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BCMA-PET
Record Dates: First submitted 2025-09-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma (MM)
Keywords: Multiple Myeloma; PET/CT; BCMA
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA and FDG (Experimental): All enrolled patients will undergo both 68Ga-BCMA nanobody PET/CT imaging and 18F-FDG PET/CT imaging.On the day of the examination (fasting is not required), an intravenous injection of the 68Ga-NOTA-BCMA nanobody will be administered, followed by PET/CT imaging approximately 0.5 to 1 hour later. Within 1 to 2 weeks, 18F-FDG PET/CT imaging will be performed, which requires an intravenous injection of 18F-FDG (fasting for at least 4 hours is required) followed by PET/CT imaging approximately 1 hour later.
  Interventions: Diagnostic Test: 68Ga-BCMA nanobody PET/CT; Diagnostic Test: 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-BCMA nanobody PET/CT — On the day of the examination (fasting is not required), an intravenous injection of the 68Ga-NOTA-BCMA nanobody will be administered, followed by PET/CT imaging approximately 0.5 to 1 hour later.
Diagnostic Test: 18F-FDG PET/CT — Within 1 to 2 weeks, 18F-FDG PET/CT imaging will be performed, which requires an intravenous injection of 18F-FDG (fasting for at least 4 hours is required) followed by PET/CT imaging approximately 1 hour later.

SUMMARY:
This study intends to employ 68Ga-NOTA-BCMA nanobody PET/CT imaging in patients with multiple myeloma to evaluate the feasibility of this technique for myeloma assessment, analyze the correlation between 68Ga-NOTA-BCMA nanobody uptake intensity and disease staging, tumor burden, and prognosis, explore its value in assessing treatment response and predicting early relapse, and compare its detection rate for myeloma lesions with that of 18F-FDG PET/CT. The results of this study may provide a more sensitive and specific imaging diagnostic method for patients with multiple myeloma and offer a basis for the individualized selection of future BCMA-targeted therapies. This study has been approved by the Ethics Committee of Peking Union Medical College Hospital.

DETAILED DESCRIPTION:
Multiple myeloma is a malignant plasma cell disorder. Real-time dynamic monitoring of the development, progression, and treatment response of myeloma remains an unmet clinical need. The development of a novel non-invasive in vivo detection technique is essential and holds significant importance for improving the prognosis of myeloma patients. Nuclear medicine plays a crucial role in the diagnosis, staging, treatment, and follow-up of multiple myeloma. The commonly used clinical nuclear imaging method, 18F-FDG PET/CT, has certain limitations in detecting myeloma lesions. B-cell maturation antigen (BCMA) is a target that is highly and specifically expressed on the surface of myeloma cells. The 68Ga-labeled nanobody targeting BCMA demonstrates high specificity in detecting myeloma lesions. Compared to traditional antibody-based probes, it offers advantages such as a simpler structure, lower molecular weight, and higher stability, showing promise as a novel non-invasive molecular imaging technique for myeloma evaluation and guiding individualized treatment. Our research group has completed the preparation, labeling, and quality control of the 68Ga-NOTA-BCMA nanobody molecular probe, as well as preclinical studies on its pharmacokinetics, pharmacodynamics, and safety evaluation.In this prospective study, patients diagnosed with multiple myeloma were enrolled to undergo 68Ga-BCMA nanobody imaging before treatment, followed by a repeat scan after treatment, to analyze its detection rate and correlation with clinical tumor burden.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed MM patients
* Written informed consent obtained and capable of undergoing follow-up.

Exclusion Criteria:

* Severely abnormal liver and kidney function
* Women who are planning pregnancy, are pregnant, or are breastfeeding, as well as those with childcare plans during the study period; subjects of childbearing potential must use effective contraceptive measures throughout the study.
* Individuals unable to lie flat for 30 minutes.
* Individuals who decline to participate in this clinical study.
* Patients with claustrophobia or other psychiatric disorders, or poor compliance that may compromise their ability to cooperate with the study procedures.
* Other circumstances deemed by the investigator as unsuitable for participation in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of 68Ga-BCMA nanobody PET/CT | through study completion, an average of 1 year
  The number of patients with positive BCMA PET results was counted and divided by the total number of individuals who completed BCMA PET imaging to calculate the detection rate of BCMA PET.

SECONDARY OUTCOMES:
Survival | through study completion, an average of 1 year
  The time to progression (TTP) in follow-up patients was analyzed using the log-rank test for survival analysis to examine the association between baseline BCMA PET positivity and TTP.

CONTACTS AND LOCATIONS:
Overall Officials: Yaping Luo, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No